CLINICAL TRIAL: NCT06466668
Title: De Oorzaak: Impact of Environmental Noise on Sleep Quality and Stress, and the Role of Auditive Sensitivity in This
Brief Title: De Oorzaak: Citizen Science Project on the Impact of Environmental Noise
Status: Enrolling by invitation | Type: Observational
Sponsor: University Hospital, Antwerp (Other)
Collaborators: Universiteit Antwerpen (Other)
Responsible Party: Sponsor
Other Study IDs: B3002024000055
Record Dates: First submitted 2024-05-13; First posted 2024-06-20 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-03

CONDITIONS: Noise Exposure; Sleep; Hyperacusis
MeSH Terms: conditions — Hyperacusis | interventions — Polysomnography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hyperacusis: participants with hyperacusis (or an increased sensitivity to sound)
  Interventions: Diagnostic Test: Sleep study; Diagnostic Test: stress-related biomarkers and microbiome composition will be assessed using saliva samples; Diagnostic Test: Audiological tests
- No hyperacusis: participants without hyperacusis (or an increased sensitivity to sound)
  Interventions: Diagnostic Test: Sleep study; Diagnostic Test: stress-related biomarkers and microbiome composition will be assessed using saliva samples; Diagnostic Test: Audiological tests

INTERVENTIONS:
Diagnostic Test: Sleep study — All subjects will undergo a polysomnography at home
Diagnostic Test: stress-related biomarkers and microbiome composition will be assessed using saliva samples — stress and stress-related inflammatory biomarkers will be tested using saliva sample
Diagnostic Test: Audiological tests — Pure tone audiometry, Uncomfortable Loudness Levels, Distortion-Product Otoacoustic Emissions, tablet test for hyperacusis, tablet test for hearing screening

SUMMARY:
"De Oorzaak" is a large-scale citizen science project aiming to assess the impact of environmental sounds on the quality of life. This particular study is a part of a broader citizen science research project "De Oorzaak", which focuses on mapping the effects of ambient noise with high resolution and on a large scale across Flanders. The specific goal of the underlying sub study is to expand our current knowledge of how ambient noise affects sleep quality and stress.

DETAILED DESCRIPTION:
The literature identifies both factors as crucial aspects of health and quality of life that are strongly influenced by ambient noise. However, it is often complex to establish a direct connection between these factors.

Sound has a significant impact on both sleep quality and quality of life. A calm, quiet environment is essential for a good night's sleep since sounds can cause interference and induce sleep disturbances. External noise, such as traffic, neighbours or city activities, can result in sleep disturbances and fatigue. In addition, sudden, loud noises such as sirens can interrupt sleep cycles, further negatively affecting the depth and quality of sleep. Furthermore, recent research demonstrated an increase in stress biomarkers in saliva during various stress conditions, including noise pollution in urban environments, as well as disruptions to the microbiome and increases in inflammatory biomarkers in saliva due to stress. However, it is challenging to directly attribute this disruption of sleep quality and increased stress levels to noise. Research often relies on participant self-reporting. "De Oorzaak" offers a unique opportunity to link sleep quality and stress (via a medical assessment) directly to environmental noise (objectivized using a sound sensor outside the bedroom window), while correcting for participants' sensitivity to it.

In order to do so, 2400 advanced sound sensors will be installed at bedroom windows of citizens across Antwerp, Ghent and Leuven to objectivize the sound landscape in these cities. Additionally, a detailed medical assessment is employed to objectivize the impact of sound on the quality of life in a subset of 120 citizens in the city of Antwerp. The goal of this assessment is to obtain an objective evaluation of sleep quality and stress and the potential association to individual oversensitivity to sound in citizens whose bedroom is located at the street side. In order to do so, citizens will be submitted to a remote sleep study with electrodes registering brain and muscle activity to determine different sleep stages as well as the potential sound-induced disruption thereof. Additionally, saliva samples will be collected to objectivize the stress experiences by the citizen involved in this project. Finally, an audiological assessment will be performed to evaluate the dynamical range of hearing thresholds and uncomfortable levels of loudness. By assessing these parameters a comparison can be made between citizens with and without hyperacusis (i.e. intolerance for daily sounds), subsequently it will be assessed whether this "sound sensitivity" results in a difference in sleep quality and stress.

ELIGIBILITY:
Inclusion Criteria:

* Adults (age 18 years old and above)
* Both male and female citizens
* Living in Antwerp
* Bedroom window allows positioning of sound sensor
* Indicated in preliminary questionnaires to be interested and willing to participate in the medical trajectory medical trajectory (i.e. sleep study, saliva sample and audiological testing)
* Equal distribution between citizens reporting both increased as decreased nuisance due to ambient noise ambient noise
* Equal distribution of participants reporting a high or low impact on their sleep quality due to Equal distribution of participants reporting a high or low impact on their sleep quality due to nighttime environmental noise

Exclusion Criteria:

* Known chronic medical conditions
* Smoking
* Bad self-reported health condition
* Diagnosed chronic diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healty population representing the citizens of Antwerp with an equal distribution between those with and without increased sensitivity to ambient noise.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-04-29 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Sound-induced sleep disturbances | Single time point (before December 31 2025)
  Polysomnographic analysis of the sleep to incedence of (micro)arousals. Using a class I sound sensor it will be assessed whether and which sounds are present at the time of these arousals.

SECONDARY OUTCOMES:
Differences in the levels of stress-related biomarkers in saliva | Single time point before sleep analysis
  Quantification of hormones (e.g., cortisol) and cytokines (e.g., IL-8) by ELISA
Differences in salivary microbiome composition | Single time point before sleep analysis
  Amplicon sequencing with the Illumina MiSeq

CONTACTS AND LOCATIONS:
Locations (1):
- Antwerp University Hospital (UZA), Edegem, Belgium

IPD SHARING:
Plan to Share IPD: Undecided